CLINICAL TRIAL: NCT06431880
Title: External Oblique Intercostal Plane Block Versus Thoracic Paravertebral Block for Post Thoracotomy Pain: A Randomized Non-inferiority Trial
Brief Title: External Oblique Intercostal Plane Block Versus Thoracic Paravertebral Block for Post Thoracotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36246PR638/4/24
Record Dates: First submitted 2024-05-16; First posted 2024-05-29 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: External Oblique Intercostal Plane Block; Thoracic Paravertebral Block; Post Thoracotomy Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External oblique intercostal plane block (Experimental): Patients will receive external oblique intercostal plane block.
  Interventions: Other: External oblique intercostal plane block
- Thoracic paravertebral block (Experimental): Patients will receive thoracic paravertebral block.
  Interventions: Other: Thoracic paravertebral block

INTERVENTIONS:
Other: External oblique intercostal plane block — Patients will receive external oblique intercostal plane block
  Arms: External oblique intercostal plane block
Other: Thoracic paravertebral block — Patients will receive thoracic paravertebral block
  Arms: Thoracic paravertebral block

SUMMARY:
The aim of this study is to compare the effectiveness of analgesia achieved by external oblique intercostal plane block (EOIPB)and thoracic paravertebral block (TPVB) for postoperative pain management in patients undergoing open thoracotomy.

DETAILED DESCRIPTION:
Acute thoracotomy pain is multifactorial in nature. It involves nociceptive and neuropathic mechanisms originating from somatic and visceral afferents. The main sources of pain are intercostal nerves, the vagus nerve and phrenic nerve in the pleura, the superficial cervical plexus, and the brachial plexus in the ipsilateral shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-III.
* Scheduled for open thoracotomy

Exclusion Criteria:

* Patients with neurological or intellectual disability.
* Infection at the injection site.
* Opioid addiction.
* Allergic reaction to local anesthetics.
* Coagulation abnormalities.
* Drug abuse.
* Pregnancy.
* Severe liver and/or renal failure.
* Uncontrolled hypertension.
* Severe cardiovascular problems.
* Diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 2 mg bolus if the numeric rating scale (NRS) > 3 to be repeated after 30 min if pain persists until the numeric rating scale < 4. numeric rating scale will be assessed at 0, 4, 8, 12, 18 and 24h postoperatively.

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperative
  Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).
Mean arterial pressure | Till the end of surgery
  Mean arterial pressure will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.
Heart rate | Till the end of surgery
  Heart rate will be recorded preoperative, before performing of block, and every 15 min till the end of surgery.
Time to the 1st rescue analgesia | 24 hours postoperatively
  All patients will receive paracetamol 1 gm every 6 h as routine analgesia. Rescue analgesia of morphine will be given as 2 mg bolus if the numeric rating scale > 3 to be repeated after 30 min if pain persists until the numeric rating scale < 4. NRS will be assessed at 0, 4, 8, 12, 18 and 24h postoperatively
Degree of pain | 24 hours postoperatively
  Degree of pain will be measured using numeric rating scale (NRS) (0 represents "no pain" while 10 represents "the worst pain imaginable").NRS will be assessed at 0, 4, 8, 12, 18 and 24h postoperatively.
Complications | 24 hour postoperatively
  Complications such as bradycardia, hypotension, nausea, vomiting, respiratory depression, local anesthetic systemic toxicity (LAST) or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, El-Gharbia Governorate, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.